CLINICAL TRIAL: NCT06525272
Title: A Phase 1 Randomized, Double-Blind, Multicenter Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of OsrhCT Administered Intrathoracically in Single and Multiple Doses in Patients With Pleurisy
Brief Title: A Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of OsrhCT in Patients With Pleurisy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Healthgen Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HY1005-2023-2-P1
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Pleurisy
Keywords: OsrhCT; Recombinant Human Chymotrypsin
MeSH Terms: conditions — Pleurisy

STUDY DESIGN:
Intervention Model Description: The study comprises two parts: Single Ascending Dose (SAD)，There are six dose groups (2000U, 4000U, 8000U, 12000U, 16000U, 20000U) and Multiple Ascending Dose (MAD),There are three dose groups (Low (TBD),Medium (TBD),High (TBD) ) both employing a multicenter, randomized, double-blind, and placebo-controlled design. Per dose group (6 receiving intrathoracic injection of OsrhCT and 2 receiving intrathoracic injection of placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double (Participant,Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Chymotrypsin(OsrhCT) (Experimental): Recombinant Human Chymotrypsin (OsrhCT), freeze-dried powder, 4,000U/vial
  Single Ascending Dose (SAD) Study:
  20ml of the prepared drug will be injected into the thoracic cavity through a chest tube.There are six dose groups (2000U, 4000U, 8000U, 12000U, 16000U, 20000U),each subject can only receive administration in one dose group, and repeated administration is not allowed.
  Multiple Ascending Dose (MAD) Study:
  20ml of the prepared drug will be injected into the thoracic cavity through a chest tube.three dose groups (low, medium, and high) will be selected for multiple dosing. Each subject will receive only one dose group and no repeat dosing.
  Interventions: Drug: Recombinant Human Chymotrypsin(OsrhCT)
- Placebo for Recombinant Human Chymotrypsin (Placebo Comparator): Placebo for Recombinant Human Chymotrypsin (OsrhCT), freeze-dried powder
  Single Ascending Dose (SAD) Study:
  20ml of the prepared drug will be injected into the thoracic cavity through a chest tube.There are six dose groups ,each subject can only receive administration in one dose group, and repeated administration is not allowed.
  Multiple Ascending Dose (MAD) Study:
  20ml of the prepared drug will be injected into the thoracic cavity through a chest tube.three dose groups (low, medium, and high) will be selected for multiple dosing. Each subject will receive only one dose group and no repeat dosing.
  Interventions: Drug: Placebo for Recombinant Human Chymotrypsin(OsrhCT)

INTERVENTIONS:
Drug: Recombinant Human Chymotrypsin(OsrhCT) — Recombinant Human Chymotrypsin (OsrhCT), provided by Wuhan Healthgen Biotechnology Corporation, 4,000U/vial, freeze-dried powder, 20ml of the prepared drug will be injected into the thoracic cavity through a chest tube.
  Other Names: Freeze-dried Powder of Recombinant Human Chymotrypsin(OsrhCT)
  Arms: Recombinant Human Chymotrypsin(OsrhCT)
Drug: Placebo for Recombinant Human Chymotrypsin(OsrhCT) — Placebo for Recombinant Human Chymotrypsin (OsrhCT), provided by Wuhan Healthgen Biotechnology Corporation, freeze-dried powder, stored at 2-8°C.
  Other Names: Freeze-dried Powder of Placebo for Recombinant Human Chymotrypsin(OsrhCT)
  Arms: Placebo for Recombinant Human Chymotrypsin

SUMMARY:
Primary Objectives:

To evaluate the safety and tolerability of single and multiple ascending doses of OsrhCT administered intrathoracically in patients with pleurisy, and to explore the DLT, MTD, and recommended effective dose of OsrhCT.

Secondary Objectives:

To evaluate the preliminary efficacy of single and multiple intrathoracic doses of OsrhCT.

Population:

Patients diagnosed with pleurisy requiring chest tube drainage.

Investigational Products:

Investigational Drug: Recombinant Human Chymotrypsin (OsrhCT), provided by Wuhan Healthgen Biotechnology Corporation, 4,000U/vial, freeze-dried powder, stored at 2-8°C.

Placebo:

Placebo for Recombinant Human Chymotrypsin (OsrhCT), provided by Wuhan Healthgen Biotechnology Corporation, freeze-dried powder, stored at 2-8°C.

Study Design:

The study comprises two parts: Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD), both employing a multicenter, randomized, double-blind, and placebo-controlled design.

Sample Size:

A total of 72 subjects (both male and female) are expected to be enrolled in this trial, including 48 subjects for single-dose administration and 24 subjects for multiple-dose administration.

DETAILED DESCRIPTION:
Primary Objectives:

To evaluate the safety and tolerability of single and multiple ascending doses of OsrhCT administered intrathoracically in patients with pleurisy, and to explore the DLT, MTD, and recommended effective dose of OsrhCT.

Secondary Objectives:

To evaluate the preliminary efficacy of single and multiple intrathoracic doses of OsrhCT.

Population:

Patients diagnosed with pleurisy requiring chest tube drainage.

Investigational Products:

Investigational Drug: Recombinant Human Chymotrypsin (OsrhCT), provided by Wuhan Healthgen Biotechnology Corporation, 4,000U/vial, freeze-dried powder, stored at 2-8°C.

Placebo:

Placebo for Recombinant Human Chymotrypsin (OsrhCT), provided by Wuhan Healthgen Biotechnology Corporation, freeze-dried powder, stored at 2-8°C.

Indication:

Pleurisy

Sample Size:

A total of 72 subjects (both male and female) are expected to be enrolled in this trial, including 48 subjects for single-dose administration and 24 subjects for multiple-dose administration.

Study Design:

The study comprises two parts: Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD), both employing a multicenter, randomized, double-blind, and placebo-controlled design.

Single Ascending Dose (SAD) Study:

Eligible pleurisy patients will receive a single intrathoracic injection of different doses of OsrhCT to evaluate safety and tolerability. There are six dose groups (2000U, 4000U, 8000U, 12000U, 16000U, 20000U). If the previous dose group shows good tolerance and safety, the next dose group will be enrolled.

The plan is to enroll 48 subjects in this phase, with 8 subjects per dose group (6 receiving intrathoracic injection of OsrhCT and 2 receiving intrathoracic injection of placebo). Each subject can only receive administration in one dose group, and repeated administration is not allowed.

Each subject will be evaluated by the investigator based on their condition during the screening process to determine the necessity of chest tube drainage or confirm their current use of a chest tube drainage. Subsequently, the investigational drug will be administered into the pleural cavity following a baseline chest X-ray. After administration, the chest tube will be clamped for 6 hours. After 6 hours, the chest tube will be opened for drainage. Subjects are allowed to clamp the drainage tube for sleeping or going out for examination. The drainage of pleural effusion will be recorded in detail. Safety checks will be performed on Day 2, and a comprehensive safety check will be performed on Day 7. Subjects will be discharged from the study if the investigator evaluates that there are no drug-related safety issues. The administration of fibrinolytic agents into the pleural cavity is prohibited before Day 7.

Multiple Ascending Dose (MAD) Study:

Eligible pleurisy patients will receive multiple intrathoracic injections of different doses of OsrhCT to evaluate safety, tolerability, and preliminary efficacy. Based on the tolerability results from the SAD study, three dose groups (low, medium, and high) will be selected for multiple dosing. Each subject will receive only one dose group and no repeat dosing. If the previous dose group shows good tolerance and safety, the next dose group will be enrolled.

The plan is to enroll 24 subjects in this phase, with 6 subjects per dose group receiving OsrhCT and 2 subjects receiving placebo. Each subject will receive the drug once daily for three consecutive days.

Each subject will be evaluated by the investigator based on their condition during the screening process to determine the necessity of chest tube drainage or confirm their current use of a chest tube drainage. Subsequently, the investigational drug will be administered into the pleural cavity following a baseline chest X-ray. The drug is administered once a day for up to 3 days, and the interval between the two administrations is 24h±1h. If pleural effusion is completely resolved before the third dose, early termination of drug administration is allowed, and the subject can enter the follow-up period. After each administration, the chest tube will be clamped for 6 hours. After 6 hours, the chest tube will be opened for drainage. Subjects are allowed to clamp the drainage tube for sleeping or going out for examination. The drainage of pleural effusion will be recorded in detail. After the last dose, subjects will be observed in the hospital for at least 4 days. Comprehensive safety checks will be performed on Day 7 and Day 30. Subjects will be discharged from the study at Day 30 if there is no safety problem as evaluated by the investigator. The administration of fibrinolytic agents into the pleural cavity is prohibited before Day 7.

Dosing Plan:

Investigational drug preparation: Dissolve the corresponding dose of the investigational drug in 20ml of normal saline for later use.All subjects will undergo chest tube drainage before the investigational drug administration. For subjects who meet the enrollment conditions, 20ml of the prepared drug will be injected into the thoracic cavity through a chest tube. After the injection is completed, the tube will be flushed with 5ml of normal saline, and then the chest tube will be clamped. Subjects will be advised to change positions to ensure adequate drug contact with the pleura (position changes are not mandatory).

Outcome Measures:

Safety Outcome Measures:

AE and SAE; Physical examination; Vital signs; Laboratory tests (complete blood count, blood biochemistry, coagulation function, and urinalysis); 12-lead ECG.

Efficacy Outcome Measures:

Changes in pleural opacity area on chest X-ray (measured as the absolute change from baseline in the percentage of pleural opacity area in the ipsilateral half of the chest on chest X-ray from pre-administration to Day 7); Relative change in pleural opacity area on chest X-ray (measured as the percentage reduction of the baseline area from pre-administration to Day 7); Drainage of pleural effusion from the first administration to Day 7; Changes in inflammatory markers (white blood cell count and C-reactive protein) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with signed informed consent;
2. Aged 18-65 years (inclusive), male or female;
3. Clinical diagnosis of pleurisy (parapneumonic pleural effusion, empyema, tuberculous pleurisy, etc.);
4. Patients with pleural effusion confirmed by chest ultrasound or CT examination and requiring chest tube drainage as assessed by the study physician, and the ultrasound report or CT image within one month shows that there are fibrous bands or encapsulated or septated effusions in the thoracic cavity;
5. Patients who cannot be fully drained after open drainage for ≥ 3 hours after chest tube drainage and meet the following conditions: The maximum depth of pleural effusion detected by ultrasound is ≥ 2 cm;
6. Women of childbearing potential must agree to use contraception (such as intrauterine device, contraceptive pills or condoms) during the study and within 3 months after the end of the study; men must agree to use effective contraception during the study and within 3 months after the end of study period.

Exclusion Criteria:

1. Known allergy to the investigational drug or its excipients;
2. Known or clinically highly suspected malignant pleural effusion;
3. Received intrathoracic injection of fibrinolytic drugs (such as urokinase, streptokinase, and alteplase) within 1 month prior to enrollment;
4. History of lung resection surgery on the same side as the chest tube drainage;
5. Evidence of abdominal lesions (e.g., pancreatic cyst or renal cyst) communicating with the pleura;
6. Currently using systemic corticosteroids and unable to discontinue;
7. HIV antibody positive;
8. History of organ transplantation;
9. Severe cardiovascular, cerebrovascular, hematologic diseases, or malignancies;
10. Abnormal laboratory values: hemoglobin <80g/L, total bilirubin >2×ULN (upper limit of normal), ALT >2.5×ULN, AST >2.5×ULN, creatinine >2×ULN; coagulation function APTT >1.5×ULN, or INR >1.5;
11. Pregnant or breastfeeding women;
12. Subjects who have participated in any drug clinical trial and received treatment within the last 3 months (excluding diagnostic skin test);
13. Any other conditions deemed unsuitable for the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety Outcome Measures | Single Ascending Dose (SAD) Study:7days;Multiple Ascending Dose (MAD) Study:30days
  Incidence of AE

SECONDARY OUTCOMES:
Efficacy Outcome Measures:Changes in pleural opacity area on chest X-ray | 7 days
  Measured as the absolute change from baseline in the percentage of pleural opacity area in the ipsilateral half of the chest on chest X-ray from pre-administration to Day 7
Efficacy Outcome Measures:Relative change in pleural opacity area on chest X-ray | 7 days
  Relative change in pleural opacity area on chest X-ray (measured as the percentage reduction of the baseline area from pre-administration to Day 7)
Efficacy Outcome Measures:Drainage of pleural effusion | 7 days
  Drainage of pleural effusion from the first administration to Day 7
Efficacy Outcome Measures:Changes in inflammatory markers | 7 days
  White blood cell count and C-reactive protein before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, MD, Principal Investigator — Shenzhen Third People's Hospital
Locations (4):
- China (4):
  - Anhui Chest Hospital, Hefei, Anhui
  - Shenzhen Third People's Hospital, Shenzhen, Guangdong
  - Wuhan Pulmonary Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No